CLINICAL TRIAL: NCT03887221
Title: A Phase I, Pharmacokinetics, Safety and Tolerability Study of Single and Multiple Oral Doses of Safinamide in Healthy Adult Chinese Volunteers
Brief Title: A Single and Multiple Dose Study to Assess How the Drug Enters, Moves Through and Exits the Body, Safety and Tolerability of Safinamide in Healthy Adult Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z7219J03
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Pharmacokinetic; Safety; Tolerability; Healthy Chinese subjects
MeSH Terms: interventions — safinamide

STUDY DESIGN:
Intervention Model Description: There will be 2 treatment groups. A total of 24 subjects will be randomized to receive 50mg or 100 mg Safinamide in Period 1 (Day 1) and Period 2 (Days 8 to 14) separated by a 7 days washout period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safinamide 50mg (Experimental): The subjects will receive 50mg safinamide on Day 1 of Period 1 and on Days 8 to 14 in period 2.
  Interventions: Drug: Safinamide 50 mg
- Safinamide 100mg (Experimental): The subjects will receive 100mg safinamide on Day 1 of Period 1 and on Days 8 to 14 in period 2.
  Interventions: Drug: Safinamide 100mg

INTERVENTIONS:
Drug: Safinamide 50 mg — Safinamide 50mg film-coated tablets will be administered to subjects in Cohort 1. The subjects will receive the tablets orally in the morning, at 8:00±1hour, under fasting conditions, with 240 mL (total volume) of still mineral water. A mouth-and-hand check will be performed immediately after dosing to ensure treatment compliance.
  Arms: Safinamide 50mg
Drug: Safinamide 100mg — Safinamide 100mg film-coated tablets will be administered to subjects in Cohort 2. The subjects will receive the tablets orally in the morning, at 8:00±1hour, under fasting conditions, with 240 mL (total volume) of still mineral water. A mouth-and-hand check will be performed immediately after dosing to ensure treatment compliance.
  Arms: Safinamide 100mg

SUMMARY:
This is a Phase I, single center, single and multiple-dose, open-label, randomised, parallel-group, pharmacokinetics, safety and tolerability study. The subjects will be randomised into two study cohorts to receive single and multiple doses of 50 mg safinamide (cohort 1), or single and multiple doses of 100 mg safinamide (cohort 2) as follows:

Cohort 1: One safinamide 50 mg film-coated tablet will be administered on day 1 followed by 7 safinamide 50 mg film-coated tablets in total from day 8 to day 14 and hence administered 1 tablet orally from day 8 to day 14.

Cohort 2: One safinamide 100 mg film-coated tablet will be administered on day 1 followed by 7 safinamide 100 mg film-coated tablets in total from day 8 to day 14 and hence administered 1 tablet orally from day 8 to day 14.

The investigational products will be administered in the morning, at 8:00±1hour, under fasting conditions, with 240 mL (total volume) of still mineral water. A mouth-and-hand check will be performed immediately after dosing to ensure treatment compliance.

The primary endpoint will assess the pharmacokinetic parameters after single and multiple dose administration of the study drug. The secondary endpoint will provide the safety and tolerability data after single and multiple dose administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: males and females, 18-45-year old inclusive
3. Ethnicity: Chinese
4. Weight: body weight ≥ 50 kg;
5. Body Mass Index: 19-26 kg/m2 inclusive
6. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting/supine position
7. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
8. No nicotine addiction (smoker subjects only): ability to abstain for smoking for the duration of the clinical study
9. Contraception and fertility (women only): women of child-bearing potential must be using at least one of the following reliable methods of contraception during the study and two weeks post-dose:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner

Women of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all women, pregnancy test result must be negative at screening and day -1.

Exclusion Criteria:

1. Electrocardiogram (12-lead ECG in supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; positive result on HIV, hepatitis B (HBV) (except for vaccination), hepatitis C (HCV). Retinal degeneration, uveitis, inherited retinopathy or severe progressive diabetic retinopathy.
6. Medications: medications, including over the counter medications, herbal remedies and traditional Chinese remedies for 2 weeks before the start of the study. In particular statins and β-Hydroxy β-methylglutaryl-CoA (HMG-CoA)reductase inhibitors in the 2 weeks before the screening visit; medicinal products that are Breast Cancer Resistance Protein (BCRP) substrates; treatment with morphine or other similar opioids, whose concomitant use with Monoamine oxidase B (MAO-B) inhibitors is contraindicated, Selective serotonin reuptake inhibitors (SSRIs), Serotonin-norepinephrine reuptake inhibitors (SNRIs), tri- or tetracyclic antidepressant, tramadol, pethidine, dextromethorphan, Monoamino oxidase (MAO) inhibitors (e.g. selegiline), meperidine derivatives and antiepileptic drugs in the 4 weeks before the screening visit; treatment with any known enzyme inhibiting or inducing agent within 4 weeks preceding the screening visit. Hormonal contraceptives for women will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study
8. Blood donation: blood donations or blood components transfusion for 3 months before this study
9. Abuse drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015-2020], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes or equivalent amount of tobacco per day within 3 months prior to day-1)
10. Abuse drug test: positive result at urine drug test at screening or day-1
11. Alcohol test: positive alcohol breath test at day -1
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians; consumption of grapefruit or products containing grapefruit within 48 hours prior to the enrolment; consumption of beverages containing xanthines (e.g. coffee, tea, soda, coffee, milk, energy drinks) within 48 hours prior to the enrolment
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Med, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Pending

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center study was conducted on 24 Healthy Adult Chinese Volunteers in China from 21 Jun 2021 to 20 Aug 2021.
Pre-assignment Details: The screening period was between Day -14 and Day -2. All the study assessments were performed as per the schedule of assessments.
Groups:
- Cohort 1 (Safinamide 50mg): The subjects received 50mg single-dose of safinamide on Day 1 orally (Period 1) and later subjects received 50mg one tablet once daily orally from Days 8 to 14 (Period 2). The single-dose in Period 1 and the first dose in Period 2 were separated by a washout interval of 7 days.
- Cohort 2 (Safinamide 100mg): The subjects received 100mg single-dose of safinamide on Day 1 orally (Period 1) and later subjects received 100mg one tablet once daily orally from Days 8 to 14 (Period 2). The single-dose in Period 1 and the first dose in Period 2 were separated by a washout interval of 7 days.
Period: Overall Study
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomised set: all subjects randomised. This analysis set was used for the analysis of demographic, baseline and background characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (5.86) | 29.9 (5.38) | 30.4 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 12 | 12 | 24
  Not Chinese | 0 | 0 | 0
  Unknown | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Safinamide Plasma Concentration (Cmax)
Description: The Cmax was determined on Day 1 (after the first dose), on Day 8 (after the first multiple doses) of Safinamide.
Time Frame: Day 1 and Day 8
Population: All randomised subjects who fulfilled the study protocol requirements in terms of investigational medicinal product (IMP) intake and had evaluable pharmacokinetic (PK) data readouts, with no major deviations that might affect the PK results. This analysis set was used for the statistical analysis of the PK summaries and analyses.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
nanogram/milliliter (ng/mL)
  Day 1 | 411.5 (96.58) | 792.1 (124.0)
  Day 8 | 465.0 (86.94) | 825.3 (183.5)

2. Primary Outcome: Time Corresponding to Occurrence of Cmax (Tmax)
Description: The tmax was determined on Day 1 (after the first dose), on Day 8 (after the first multiple dose) of Safinamide.
Time Frame: Day 1 and Day 8
Population: All randomised subjects who fulfilled the study protocol requirements in terms of IMP intake and had evaluable PK data readouts, with no major deviations that might affect the PK results. This analysis set was used for the statistical analysis of the PK summaries and analyses.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour (h)
  Day 1 | 1.500 [0.50 to 3.00] | 1.750 [1.00 to 3.00]
  Day 8 | 2.000 [0.50 to 8.00] | 1.508 [1.00 to 3.00]

3. Primary Outcome: Area Under the Concentration-time Curve From Single-dose Administration to the Last Quantifiable Concentration-time t (AUC0-t)
Description: The (AUC0-t) was determined on Day 1 (after the first dose), on Day 8 (after the first multiple doses) of Safinamide.
Time Frame: Day 1 and Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour* nanogram/milliliter (h*ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour* nanogram/milliliter (h*ng/mL)
  Day 1 | 11560 (2170) | 20790 (3131)
  Day 8 | 6652 (985.5) | 12130 (1846)

4. Primary Outcome: Area Under the Concentration-time Curve in the Tau Interval (From Single Dose Administration to 24 h Post Dose) (AUC0-24h)
Description: The (AUC0-24h) was determined on Day 1 (after the first dose), on Day 8 (after the first multiple dose) of safinamide.
Time Frame: Day 1 and Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour*nanogram/milliliter (h*ng/mL)
  Day 1 | 6291 (1158) | 11420 (1727)
  Day 8 | 6649 (986.3) | 12090 (1931)

5. Primary Outcome: Last Quantifiable Concentration (Clast/Ct)
Description: The (Clast/Ct) was determined on Day 1 (after the first dose) of safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
nanogram/milliliter (ng/mL) | 23.01 (9.306) | 37.26 (7.483)

6. Primary Outcome: Terminal Elimination Rate Constant (Kel)
Description: Apparent terminal elimination rate constant, calculated, if feasible, from the slope of a log-linear regression using at least 3 last concentration > lower limit of quantification (LLOQ) points. The Kel was determined on Day 1 (after the first dose) of safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour (h) | 0.02967 (0.004188) | 0.03019 (0.002283)

7. Primary Outcome: Apparent Terminal Elimination Half Life (t1/2)
Description: Apparent terminal elimination half-life, calculated, if feasible, as ln2/Kel. The t1/2 will be determined on Day 1 (after the first dose) of Safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour (h) | 23.79 (3.391) | 23.08 (1.740)

8. Primary Outcome: Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex)
Description: The %AUCex was determined on Day 1 (after the first dose) of Safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
percentage (%) | 6.594 (2.931) | 5.672 (1.077)

9. Primary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC(0-inf))
Description: Area under the concentration-time curve extrapolated to infinity, calculated, if feasible, as AUC0-t + Ct/Kel, where Ct is the last measurable drug concentration. The AUC(0-inf) was determined on day 1 (after the first dose) of Safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour*nanogram/milliliter (h*ng/mL) | 12380 (2424) | 22030 (3290)

10. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vd/F)
Description: Apparent volume of distribution associated with the terminal slope, calculated, if feasible, as Dose/(AUC0-∞*Kel). The Vd/F was determined on Day 1 (after the first dose) of safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
milliliter (mL) | 142700 (33040) | 154800 (29600)

11. Primary Outcome: Apparent Clearance Following Oral Administration (CL/F)
Description: Apparent total body clearance, calculated, if feasible, as Dose/AUC0-∞. The CL/F was determined on Day 1 (after the first dose) of safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter/ hour (mL/h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
milliliter/ hour (mL/h) | 4159 (697.2) | 4634 (707.1)

12. Primary Outcome: Mean Residence Time (MRT)
Description: Mean residence time, calculated, if feasible, as AUMC0-∞/AUC0-∞, where AUMC0-∞ is area under the moment concentration-time curve extrapolated to infinity. The MRT was determined on Day 1 (after the first dose) of Safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour (h) | 34.65 (5.324) | 33.12 (1.988)

13. Primary Outcome: Area Under the First Moment of the Concentration-time Curve (AUMC)
Description: The AUMC was determined on Day 1 (after the first dose) of Safinamide.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour2* nanogram/milliliter (h2*ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour2* nanogram/milliliter (h2*ng/mL) | 431100 (131600) | 729400 (117100)

14. Primary Outcome: Maximum Safinamide Plasma Concentration at Steady State (Cmax_ss)
Description: The Cmax_ss was determined on day 14 (after the multiple-dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nnaogram/milliliter (ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
nnaogram/milliliter (ng/mL) | 782.8 (174.4) | 1501 (249.6)

15. Primary Outcome: Time Corresponding to Occurrence of Cmax_ss at Steady State (tmax_ss)
Description: The tmax_ss was determined on day 14 (after the multiple-dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour (h) | 2.017 [1.00 to 6.00] | 1.483 [0.50 to 4.00]

16. Primary Outcome: Minimum Observed Concentration at Steady State (Cmin_ss)
Description: The Cmin_ss was determined on day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram/liter (ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
nanogram/liter (ng/mL) | 358.3 (107.8) | 583.2 (117.2)

17. Primary Outcome: Area Under the Concentration-time Curve at Steady State From the Last Dose Administration to the Last Observed Concentration Time t (AUC0-t_ss)
Description: The AUC0-t_ss was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour*nanogram/milliliter (h*ng/mL) | 24170 (6349) | 42420 (6676)

18. Primary Outcome: AUC Over the Dosing Interval at Steady State (AUC0-τ_ss)
Description: The AUC0-τ_ss was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
hour*nanogram/milliliter (h*ng/mL) | 13150 (2781) | 23100 (3541)

19. Primary Outcome: Average Safinamide Plasma Concentration at Steady State(Cave_ss)
Description: Average safinamide plasma concentration at steady state, calculated as AUC0- 24h_ss /tau (24 h). The Cave_ss was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
nanogram/milliliter (ng/mL) | 548.0 (115.9) | 962.4 (147.5)

20. Primary Outcome: Accumulation Ratio, Based on AUC (Racc,AUC)
Description: Racc,AUC was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
ratio | 2.101 (0.2525) | 2.027 (0.1367)

21. Primary Outcome: Accumulation Ratio, Based on Cmax (Racc,Cmax)
Description: Racc,Cmax was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
ratio | 1.939 (0.3691) | 1.898 (0.1594)

22. Primary Outcome: Peak-trough Fluctuation Over One Dosing Interval at Steady-state (DF%)
Description: Peak-trough fluctuation over one dosing interval at steady-state, calculated as (Cmax,ss - Cmin,ss)/Cave,ss*100. The DF% was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
percentage (%) | 77.75 (13.42) | 95.17 (11.90)

23. Primary Outcome: Apparent Volume of Distribution at Steady-state Associated With the Terminal Slope (Vd/F_ss)
Description: Apparent volume of distribution at steady-state associated with the terminal slope, calculated, if feasible, as Dose/( AUC0-24h_ss*Kel). The Vd/F_ss was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
milliliter (mL) | 134400 (28640) | 153100 (30250)

24. Primary Outcome: Apparent Total Body Clearance at Steady-state, (CL/F_ss)
Description: The CL/F_ss was determined on Day 14 (after the multiple dose) of Safinamide.
Time Frame: Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter/hour (mL/h)
Arm/Group | Cohort 1 (Safinamide 50mg) | Cohort 2 (Safinamide 100mg)
Number analyzed (Participants) | 11 | 12
milliliter/hour (mL/h) | 3933 (705.8) | 4426 (692.0)

25. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Safety and general tolerability were assessed for safinamide.
Time Frame: Day 1 to18
Population: All randomised subjects who receive at least one dose of the investigational medicinal product(s). This analysis set will be used for the safety analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (Safinamide 50mg) Single Dose: The subjects received 50mg single-dose of safinamide on Day 1 orally (Period 1).
- Cohort 2 (Safinamide 100mg) Single Dose: The subjects received 100mg single-dose of safinamide on Day 1 orally (Period 1).
- Cohort 1 (Safinamide 50mg) Multiple Dose: The received 50mg one tablet once daily orally from Days 8 to 14 (Period 2).
- Cohort 2 (Safinamide 100mg) Multiple Dose: The received 100mg one tablet once daily orally from Days 8 to 14 (Period 2).
Arm/Group | Cohort 1 (Safinamide 50mg) Single Dose | Cohort 2 (Safinamide 100mg) Single Dose | Cohort 1 (Safinamide 50mg) Multiple Dose | Cohort 2 (Safinamide 100mg) Multiple Dose
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  TEAE | 6 | 7 | 5 | 4
  TEAE Related to IMP | 6 | 7 | 5 | 4

ADVERSE EVENTS:
Time Frame: From Screening to final visit/ Early termination visit (Day 18)
Groups:
- Cohort 1 (Safinamide 50mg) Multiple Dose: The subjects received 50mg one tablet once daily orally from Days 8 to 14 (Period 2).
- Cohort 2 (Safinamide 100mg) Multiple Dose: The subjects received 100mg one tablet once daily orally from Days 8 to 14 (Period 2).
Arm/Group | Cohort 1 (Safinamide 50mg) Single Dose | Cohort 2 (Safinamide 100mg) Single Dose | Cohort 1 (Safinamide 50mg) Multiple Dose | Cohort 2 (Safinamide 100mg) Multiple Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 7/12 | 5/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Safinamide 50mg) Single Dose (N=12) | Cohort 2 (Safinamide 100mg) Single Dose (N=12) | Cohort 1 (Safinamide 50mg) Multiple Dose (N=12) | Cohort 2 (Safinamide 100mg) Multiple Dose (N=12)
Somnolence (Nervous system disorders) | 3 (3) | 5 (5) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains confidential information of Zambon S.p.A., Italy. Do not copy or distribute without written permission from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT03887221/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT03887221/SAP_001.pdf